CLINICAL TRIAL: NCT05802992
Title: A Single-center Clinical Trial to Evaluate the Efficacy and Safety of Colchicine Combined With Conventional Therapy in Multiple Myeloma Patients
Brief Title: The Efficacy and Safety of Colchicine Combined With Conventional Therapy in Multiple Myeloma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Hongming Huang, Deputy Director of Hematology Department, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K043-01
Record Dates: First submitted 2023-03-03; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Colchicine
MeSH Terms: conditions — Multiple Myeloma | interventions — Colchicine; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will be treated with colchicine, lenalidomide and dexamethasone, every 28 days as a cycle.
  Interventions: Drug: Colchicine; Drug: Lenalidomide
- Control group (Active Comparator): Patients will receive lenalidomide and dexamethasone as background treatment, every 28 days as a cycle.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Colchicine — The investigational drug colchicine was used at a daily dose of 0.5-1 mg. In every cycle, lenalidomide was administered at 10-25 mg (days 1-21). Dexamethasone 40mg (≤75 years old) or 20mg (>75 years old) per week.If the weekly dose of dexamethasone is 40mg, it should be taken in the first two days of the week, 20mg per day; If the weekly dose is 20mg or take the lower dose on the first day of each week.
  If the patient needs to be treated with the investigational drug colchicine on the day of dexamethasone administration, he should take dexamethasone orally within 3 hours before the administration of colchicine.
  Other Names: Lenalidomide; Dexamethasone
  Arms: Experimental group
Drug: Lenalidomide — In every cycle, lenalidomide was administered at 10-25 mg (days 1-21). Dexamethasone 40mg (≤75 years old) or 20mg (>75 years old) per week.If the weekly dose of dexamethasone is 40mg, it should be taken in the first two days of the week, 20mg per day; If the weekly dose is 20mg or take the lower dose on the first day of each week.
  Other Names: Dexamethasone

SUMMARY:
To evaluate the efficacy and safety of investigational drug Colchicine combined with conventional lenalidomide based therapy in multiple myeloma subjects who had received first-line therapy (including Chimeric antigen receptor T-Cell immunotherapy (CART) treatment), and to evaluate the quality of life of the patients.

DETAILED DESCRIPTION:
This study is expected to be carried out from March 2022 to December 2024. About 30 patients with multiple myeloma who have received at least first-line of treatment (including Chimeric antigen receptor T-Cell immunotherapy (CART) treatment) will be randomly assigned to the experimental group or the control group at 2:1. By comparing the relevant data such as efficacy evaluation and safety evaluation after treatment, the principal investigator will write and publish the paper.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of multiple myeloma Have received at least one-line treatment Must be able to swallow tablets

Exclusion Criteria:

Resistance to or intolerance to therapeutic agents such as bortezomib or lenalidomide Allergy to the experimental drug or its ingredients Has invaded the central nervous system Severe cardiovascular, liver and kidney failure, severe chronic obstructive pulmonary disease (COPD), and moderate to severe asthma Active hepatitis B or C infection HIV seropositivity Is participating in other clinical trials or has participated in other clinical trials within the past two weeks Other factors that the researchers determined were not suitable for the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum M protein | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of Serum M protein before and after treatment
Proportion of bone marrow plasma cells | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the proportion of bone marrow plasma cells before and after treatment
Serum protein electrophoresis (SPEP) and urine protein electrophoresis (UPEP） | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of SPEP and UPEP before and after treatment
Serum free light chain (FLC) | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of Serum FLC before and after treatment

SECONDARY OUTCOMES:
Imaging（X ray/CT/MRI） | [Time Frame:Baseline, at the end of every two cycles (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of Serum M protein before and after treatment
Complete blood count (CBC) | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of CBC before and after treatment
Blood biochemistries | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the level of Serum M protein before and after treatment
Eastern Cooperative Oncology Group (ECOG) Score | [Time Frame:Baseline, at the end of each cycle (each cycle is 35 days). From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months]
  Changes of the ECOG score before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongming Huang, PhD, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Not planning sharing at present.

REFERENCES:
- [Background] Dasgeb B, Kornreich D, McGuinn K, Okon L, Brownell I, Sackett DL. Colchicine: an ancient drug with novel applications. Br J Dermatol. 2018 Feb;178(2):350-356. doi: 10.1111/bjd.15896. Epub 2018 Jan 3. PMID 28832953
- [Background] Cho JH, Joo YH, Shin EY, Park EJ, Kim MS. Anticancer Effects of Colchicine on Hypopharyngeal Cancer. Anticancer Res. 2017 Nov;37(11):6269-6280. doi: 10.21873/anticanres.12078. PMID 29061810
- [Background] Zhang T, Chen W, Jiang X, Liu L, Wei K, Du H, Wang H, Li J. Anticancer effects and underlying mechanism of Colchicine on human gastric cancer cell lines in vitro and in vivo. Biosci Rep. 2019 Jan 15;39(1):BSR20181802. doi: 10.1042/BSR20181802. Print 2019 Jan 31. PMID 30429232
- [Background] Bell CJ, Potts KG, Hitt MM, Pink D, Tuszynski JA, Lewis JD. Novel colchicine derivative CR42-24 demonstrates potent anti-tumor activity in urothelial carcinoma. Cancer Lett. 2022 Feb 1;526:168-179. doi: 10.1016/j.canlet.2021.11.028. Epub 2021 Nov 25. PMID 34838691
- [Background] Livneh A, Zemer D, Langevitz P, Shemer J, Sohar E, Pras M. Colchicine in the treatment of AA and AL amyloidosis. Semin Arthritis Rheum. 1993 Dec;23(3):206-14. doi: 10.1016/s0049-0172(05)80042-3. PMID 8122124
- [Background] JYO T, ENDOH H. [Clinical experience with Colcemid in true polycythemia and chronic myelogenic leukemia]. Naika Hokan. 1961 Jul 20;8:607-15. No abstract available. Japanese. PMID 13791163
- [Background] Urbaniak A, Jousheghany F, Pina-Oviedo S, Yuan Y, Majcher-Uchanska U, Klejborowska G, Moorjani A, Monzavi-Karbassi B, Huczynski A, Chambers TC. Carbamate derivatives of colchicine show potent activity towards primary acute lymphoblastic leukemia and primary breast cancer cells-in vitro and ex vivo study. J Biochem Mol Toxicol. 2020 Jun;34(6):e22487. doi: 10.1002/jbt.22487. Epub 2020 Mar 5. PMID 32141170